CLINICAL TRIAL: NCT07221760
Title: An Open-label Single Center, Single Participant Study of an Experimental Antisense Oligonucleotide Treatment for Dentatorubral-pallidoluysian Atrophy (DRPLA) Due to ATN1 Mutation
Brief Title: Personalized Antisense Oligonucleotide for A Single Participant (nL62541) With ATN1 Gene Mutation
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: n-Lorem Foundation (Other)
Collaborators: Dell Children's Medical Center of Central Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007386
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Dentatorubral-Pallidoluysian Atrophy
MeSH Terms: conditions — Myoclonic Epilepsies, Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: nL-ATN1-001

INTERVENTIONS:
Drug: nL-ATN1-001 — Personalized Antisense Oligonucleotide

SUMMARY:
This research project entails delivery of a personalized antisense oligonucleotide (ASO) drug designed for a single participant with dentatorubral-pallidoluysian atrophy (DRPLA) due to a heterozygous pathogenic CAG trinucleotide expansion in ATN1

DETAILED DESCRIPTION:
This is an interventional study to evaluate the safety and efficacy of treatment with an individualized antisense oligonucleotide (ASO) treatment in a single participant with DRPLA due to a heterozygous pathogenic CAG trinucleotide expansion in ATN1

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent provided by the participant (when appropriate), and/or participant's parent(s) or legally authorized representative(s)
* Ability to travel to the study site and adhere to study-related follow-up examinations and/or procedures and provide access to participant's medical records
* Genetically confirmed Dentatorubral-pallidoluysian atrophy (DRPLA) due to ATN1 mutation

Exclusion Criteria:

* Use of investigational medication within 5 half-lives of the drug at enrolment
* Participant has any condition that in the opinion of the Site Investigator would ultimately prevent the completion of study procedures

Min Age: 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Seizures | Baseline to 24 months
  Change in seizure length from baseline to every 3 months post nL-ATN1-002 administration as measured by routine electroencephalography (EEG) (changes in frequency of ictal and interictal discharges, evoked potentials, and changes in EEG background)
Seizures | Baseline to 24 months
  Change in seizure length from baseline to every 3 months post nL-ATN1-002 administration as measured by seizure tracking (changes in number and length of seizures)
Seizures | Baseline to 24 months
  Change in seizure frequency and seizure medication use from baseline to every 3 months post nL-ATN1-002 administration as measured by seizure tracking (reported with seizure dates and use of seizure medication)

SECONDARY OUTCOMES:
Quality of Life and Caregiver Burden | Baseline to 24 months
  Change in quality of life and caregiver burden from baseline to 6-, 12-, 18-, and 24- months post nL-ATN1-002 administration as measured by the Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD)
Quality of Life and Caregiver Burden | Baseline to 24 months
  Change in quality of life and caregiver burden from baseline to 6-, 12-, 18-, and 24- months post nL-ATN1-002 administration as measured by Caregiver Global Impression of Change Questionnaire (CaGL-C)
Health Status | Baseline to 24 months
  Change in comorbities from baseline to 6-, 12-, 18-, and 24-months post nL-ARN1-002 administration as measured by the Caregiver Priorities - Comorbidities and Health Evaluation Checklist (CPCHECKlist)
Dysphagia | Baseline to 24 months
  Change in swallow function and number of aspiration pneumonias (PNAs) from baseline to 12- and 24-months post nL-ATN1-002 administration as measured by Modified Barium Swallow Study (MBSS)
Dysphagia | Baseline to 24 months
  Change in swallow function and number of aspiration pneumonias (PNAs) from baseline to 12- and 24-months post nL-ATN1-002 administration as measured by adverse events of aspiration PNAs
Incidence and Severity of Treatment Emergent Adverse Events [Safety and Tolerability] | Baseline to 24 months
Incidence of Treatment-Emergent Abnormalities in Physical and Neurological Exams [Safety and Tolerability] | Baseline to 24 months
Incidence of Treatment-Emergent Abnormalities in Safety Labs (CSF, chemistry, hematology, coagulation, and urinalysis) [Safety and Tolerability] | Baseline to 24 months

OTHER OUTCOMES:
Developmental Skills | Baseline to 24 months
  Change in developmental skills from baseline to 6-, 12-, 18-, and 24- months post nL-ATN1-002 administration as measured by Developmental Profile 4 (DP-4) (physical, adaptive behavior, social-emotional, cognitive, and communication scores)
Developmental Skills | Baseline to 24 months
  Change in developmental skills from baseline to 6-, 12-, 18-, and 24- months post nL-ATN1-002 administration as measured by Bayley Scales of Infant Development 4 (BSID-4) (cognition, communication, motor, and adaptive behavior scores)
Developmental Skills | Baseline to 24 months
  Change in developmental skills from baseline to 6-, 12-, 18-, and 24- months post nL-ATN1-002 administration as measured by Observer Reported Communication Ability (ORCA)
Ataxia | Baseline to 24 months
  Change in ataxia from baseline to 6-, 12-, 18-, and 24- months post nL-ATN1-002 administration as measured by Scale for Assessment and Rating of Ataxia (SARA)
Brain Changes | Baseline to 24 months
  Change in brain MRIs from baseline to 12- and 24- months post nL-ATN1-002 administration as measured by ventricular size on brain MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Dell Children's, Austin, Texas, United States